CLINICAL TRIAL: NCT03607318
Title: Brief Alcohol Intervention and mHealth Booster for Suicidal Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Kimberly H. McManama O'Brien, Instructor in Psychiatry, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00028139
Record Dates: First submitted 2018-05-01; First posted 2018-07-31 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Alcohol Drinking; Suicide, Attempted; Adolescent Behavior
Keywords: alcohol; suicide; adolescents
MeSH Terms: conditions — Alcohol Drinking; Suicide, Attempted; Adolescent Behavior; Suicide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iASIST (Experimental): iASIST, involves 1) an individual intervention with the adolescent in which motivational enhancement techniques are used to explore alcohol use as a risk factor for continued suicide-related thoughts and behaviors and to create a change plan, 2) a subsequent family intervention using motivational enhancement techniques to align the parent with the adolescent to strengthen the adolescent's self-efficacy and commitment to the change plan as well as the parent's ability to support the adolescent in their plan to reduce or stop drinking, and 3) a post-discharge mHealth booster to adolescents focused on strengthening their commitment to the change plan, and to parents focused on their commitment, confidence, and ability related to supporting the adolescent in reducing or stopping drinking.
  Interventions: Behavioral: iASIST
- Attention-Matched Comparison (Active Comparator): The attention-matched comparison condition involves one psychoeducation session focused on the role of a healthy lifestyle in mental health and an additional family intervention, in which the adolescent will review handouts from the session with the parent, facilitated by the interventionist. In addition, adolescents and parents assigned to the comparison will receive a post-discharge mHealth control about the maintenance of a healthy lifestyle with the same frequency and type of interaction as the iASIST mHealth booster.
  Interventions: Behavioral: iASIST

INTERVENTIONS:
Behavioral: iASIST — Integrated Alcohol and Suicide Intervention for Suicidal Teens

SUMMARY:
The primary goal of this study is to test the acceptability and feasibility of iASIST (integrated Alcohol and Suicide Intervention for Suicidal Teens), a novel adjunctive intervention for alcohol use and alcohol-related suicidal thoughts and behaviors for suicidal adolescent inpatients.

The investigators will first conduct an open trial with 10 adolescents and their parents to test iASIST and make subsequent changes to the booster. Next, the investigators will conduct a randomized trial with 50 adolescents and their parents to test the feasibility and acceptability of iASIST as well as associations with alcohol- and suicide-related outcomes at 3 months post-discharge, relative to participants who receive an attention-matched comparison condition focused on the role of a healthy lifestyle in mental health that includes a post-discharge mHealth control targeting the maintenance of a healthy lifestyle.

DETAILED DESCRIPTION:
The primary goal of this study is to test the acceptability and feasibility of iASIST (integrated Alcohol and Suicide Intervention for Suicidal Teens), a novel adjunctive intervention for alcohol use and alcohol-related suicidal thoughts and behaviors for suicidal adolescent inpatients.

The intervention in this study, iASIST (integrated Alcohol and Suicide Intervention for Suicidal Teens), involves three components: 1) an individual intervention with the adolescent in which motivational enhancement techniques are used to explore alcohol use as a risk factor for continued suicide-related thoughts and behaviors in order to build the adolescent's motivation to reduce or stop their alcohol use and to create a complementary change plan, 2) a subsequent family intervention in which the interventionist facilitates a discussion between the adolescent and parent about the change plan using motivational enhancement techniques to align the parent with the adolescent to strengthen the adolescent's self-efficacy and commitment to the change plan as well as the parent's ability to support the adolescent in their plan to reduce or stop drinking, and 3) a post-discharge mHealth booster to adolescents focused on strengthening their commitment to the change plan, and to parents focused on their commitment, confidence, and ability related to supporting the adolescent in reducing or stopping drinking. The investigators will first conduct an open trial with 10 adolescents and their parents to test iASIST and make subsequent changes to the booster. Next, the investigators will conduct a randomized trial with 50 adolescents and their parents to test the feasibility and acceptability of iASIST as well as associations with alcohol- and suicide-related outcomes at 3 months post-discharge, relative to participants who receive an attention-matched comparison condition focused on the role of a healthy lifestyle in mental health that includes a post-discharge mHealth control targeting the maintenance of a healthy lifestyle.

The investigators anticipate that adolescents who receive iASIST, relative to the comparison condition, will have increased negative alcohol expectancies, alcohol situational confidence, mental health and/or substance abuse service use, parental monitoring, parent-child communication about alcohol, and decreased frequency of alcohol use, positive alcohol expectancies, suicide ideation, plans, and attempts at 3 month follow-up. Although the investigators do not expect statistically significant differences due to the small sample size, they will calculate confidence intervals around the effect sizes. Data will be informative for designing a fully powered clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Must be currently hospitalized for suicide ideation or attempt
* Must have used alcohol in past 3 months, indicated by selecting "yes" on the screening question ["Have you drank alcohol in the past 3 months?"]
* Must be between the age of 13-17
* The adolescent and parent/guardian must own a smartphone
* Must have the ability to communicate in English.

Exclusion Criteria:

* developmental delay
* autism spectrum disorder
* psychosis

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Groups are stratified by self-identified gender
Enrollment: 40 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Alcohol Use measured by the Timeline Followback Assessment | 3 months
  frequency of alcohol use
Suicide Attempts measured by the Columbia Suicide Severity Rating Scale | 3 months
  quantity of suicide attempts
Suicide Ideation measured by the Suicide Ideation Questionnaire, Jr | 1 month
  severity of suicide ideation
Alcohol Use measured by the Timeline Followback Assessment | 3 Months
  Quantity of Alcohol Use

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States